CLINICAL TRIAL: NCT02737111
Title: How do Families Experience Receiving a Positive Diagnosis for an Inherited Cardiac Condition for a Child? The Experiences of Children With a Diagnosis, Their Parents and Siblings.
Brief Title: Families' Experiences of Paediatric ICC Diagnosis
Acronym: FEPICCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Ben Williams Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015PC002B
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Inherited Cardiac Conditions
MeSH Terms: interventions — Informed Consent; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Initial Screening Process — The doctor who meets with the family to share the diagnosis will give the participants a flyer about the research study at the end of their consultation and will briefly explain the study aim and purpose. Following this, the ICC Service Clinical Nurse Specialists (CNS) and the primary researcher will identify patients who meet the inclusion and exclusion criteria and all patients who are eligible to take part will be contact by a CNS shortly after a child receives a diagnosis to follow up with the family, and ask permission for the primary researcher to contact the child's parents to discuss the study.
Behavioral: Information and Informed Consent — The researcher will contact parents of patients who agreed some weeks after receiving the diagnosis, check inclusion criteria, and information sheets will be provided. Individuals who consent to participate will arrange to meet with the researcher in their family home or at the hospital. When they meet, the researcher will go through the participant information sheet with the individuals, and gain written consent for participation
Behavioral: Interview — Families who wish to take part will be invited to participate in an interview 2-3 months after they received the diagnosis from the hospital. At least ten families (and therefore at least 30 individuals including children with the diagnosis, parents and siblings) will be interviewed separately, about their experiences of the communication about the diagnosis to them, their child or their siblings. Younger children may do some drawings with the researcher about their experiences, and the researcher will ask questions about these drawings.Participants can be included even if not all family members wish to take part.
Behavioral: Validated Questionnaires — Each member of the family will complete the mood and quality of life questionnaires.
Behavioral: Debrief — At the end of each interview the research will explore with the individual to discuss how they found the experience and answer any questions they might have and review the questionnaires that they completed. The researcher will then meet with children and parents together to discuss the experience as a family.Information will be shared with families about options for accessing support including the paediatric psychology service at the hospital or local support services, if they wish. After the interviews, the researcher will send a letter to participants GP and medical team to inform them that they are taking part.

SUMMARY:
This study aims to further understand the experiences of children, their parents and siblings around the time when the child and their family are informed of a diagnosis of an inherited cardiac condition (ICC). The researchers are interested to understand how families experience the process of receiving a diagnosis of an ICC, and explore experiences from multiple perspectives within the family (i.e. parents, children and siblings).

The Primary Project Objective:

How do children, their parents and siblings experience the communication of a diagnosis of an inherited cardiac condition (ICC)? What is found to be helpful and less helpful?

The Secondary Project Objective:

To explore qualitatively how families experience the communication of a positive diagnosis for an inherited cardiac condition for a child and will seek the perspectives of the child with the diagnosis, their siblings and parents.

DETAILED DESCRIPTION:
Background Information and Study Rationale:

An ICC comprise of a number of conditions that affect either the heart muscle (cardiomyopathies), or the electrical circuits of the heart (ion channelopathies). ICCs can result in the heart working ineffectively, dangerous arrhythmias and sudden death. The last decade has seen dramatic advances in understanding of the pathology of ICCs. More than 50 ICCs have been recognised and genetics tests are increasingly available. Epidemiological evidence suggests a combined total prevalence for ICCs of about 340,000 in the UK.

In response to advances in medical and genetic understanding of ICCs, ICC services have also grown dramatically, accompanied by commissiioning guidelines, and when an ICC is diagnosed there are implications not only for the patient themselves but for relatives. For families affected by inherited cardiac conditions, the layers of impact can be complex. When a child receives a positive diagnosis there can be implications for parents and siblings not only of living with the child's diagnosis, but also for one's own health and wellbeing. This can lead to uncertainty about the health of others in the family and subsequent medical investigates.

To the researchers' knowledge, there is little published evidence which aims to understand the experiences of children and their siblings of the communication around their ICC condition. Therefore ICC services risk of relying on our own clinical intuition or the views of parents rather than hearing directly from children and young people themselves. This present study therefore proposed to explore qualitatively how families experience the communication of a positive diagnosis for an inherited cardiac condition for a child and will seek the perspectives of the child with the diagnosis, their siblings and parents.

Participants will be recruited from a ICC service at an NHS Hospital in London. Paedaitric patients (who have been given an ICC diagnosis) and their siblings will be aged 8-16, and their Parents. Patient recruitment at a site will only commence once the trial team has ensured that the following approval/essential documents are in place:

1. The main REC approval,
2. Final sponsorship and/or R&D approval (NHS Permission),
3. Local Site Delegation of Duties and Signature Log is completed.

All subjects who wish to enter the study will be fully screened and consented by the Chief Investigator (CI), or one of the qualified clinicians involved in the study as the Researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 8 - 16 who have received a positive diagnosis of an inherited cardiac condition from the ICC service at the hospital within the last 3 months, their parents and siblings.
2. Siblings of children who have received a diagnosis of an inherited cardiac condition who are between the ages of 8 and 16 years.
3. Children will only participate if they are already aware of their diagnosis or their sibling's diagnosis.
4. Children will only participate if they and a parent/person with parental responsibility have both consented to take part.
5. Parents will only take part if they have given informed consent

Exclusion Criteria:

1. Children who are unable to communicate verbally will not be included in the research as they would be unable to consent to their involvement in the research and alternative means of data collection would be required.

Discontinuation/ withdrawal of Pariticpants and Stopping Rules:

Participants can withdraw their participation from the study at any time without giving a reason and if this happens, the data collected from their interviews/questionnaires will not be used in the study results. Adult participants will be told that they can tell the researcher if they would like to withdraw. The researcher will agree a word or sign with child participants to indicate that they would like to stop taking part and the researcher will then ask them whether they would like the data used to be included in the results of the study.

The researcher will continue to recruit participants until there is sufficient data for qualitative analysis of interviews.

It is unlikely that the study will be stopped prematurely but this might occur if insufficient numbers of participants are able to be recruited from one or more of the patient samples (i.e. children with a diagnosis, parents or siblings) in the designated time frame.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Experience of recieving a diagnosis of an ICC. | Interviews will occur within 2-3 months of recieiving the diagnosis
  Semi-structured interviews (Child, Sibling and Parent version) will be transcriped and analysed using thematic analysis, whereby common themes will be identified within and between participant interviews. Thematic analysis is a method for identifying, analysing and reporting patterns (themes) within data. Thematic analysis is a way to organise and describe a data set from qualitative interviews in rich detail.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Till, Doctor, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
All adult participants will be invited to a presentation of the research findings and will be given the option of receiving a final summary of the research findings once the study has been written up for publication.
  All child participants will also be invited to attend a separate presentation of the findings and will be offered a child friendly summary of the results. The researcher will provide a contact email address should participants have any further questions regarding the study and/or results.
  A report of the analysis will be written and a selection of anonymised quotations/extracts demonstrating each theme will be selected to accompany the report.
  It is intended that the research will be published in a peer-reviewed journal.